CLINICAL TRIAL: NCT06924775
Title: Impact of Jump Rope Training on the Isokinetic Shoulder Profile in CrossFit Practitioners
Brief Title: Jump Rope Training and Shoulder Isokinetics in CrossFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Maximiliano Torres-Banduc, PhD., University of Americas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23/2022
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Evaluation of the Effects of Weighted Jump Rope Training on the Isokinetic Shoulder Profile in CrossFit Practitioners
Keywords: Isokinetic shoulder profile; Weighted jump rope training; Rotational peak torque; Muscle imbalance; Injury prevention; CrossFit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Weighted jump rope training group (Experimental): A progressive six-week jump rope protocol focusing on simple unders was completed three times per week, individually or in groups, before regular sessions. Training was supervised by final-year kinesiology students. Based on Duzgun et al. (2010), jumps increased weekly: Week 1-D1: 6×25, D2: 3×50, D3: 4×50 (500 total); Week 2-4×50, 4×75, 4×50 (750); Week 3-4×75, 4×75, 4×100 (1000); Week 4-6×75, 6×75, 5×70 (1250); Week 5-5×100, 4×150, 4×100 (1500); Week 6-5×150, 6×100, 4×100 (1750). Rest between sets: 1 min. Participants were advised to avoid prior intense activity, maintain steady pace, and received positive reinforcement as needed.
  Interventions: Other: Weighted jump rope training

INTERVENTIONS:
Other: Weighted jump rope training — Unlike isolated jump rope studies, this intervention was embedded within the participants' habitual CrossFit routine, enhancing ecological validity. Performing the jump rope protocol immediately prior to regular training-rather than as a stand-alone session-was intended to promote warm-up and neuromuscular priming benefits. The use of a weighted rope introduced a resistance stimulus that is rarely incorporated in jump rope interventions.

SUMMARY:
The goal of this quasi-experimental clinical trial is to evaluate whether weighted jump rope (WJR) training can improve the isokinetic shoulder strength profile in male and female CrossFit practitioners.

The main questions it aims to answer are:

* Does six weeks of WJR training affect internal and external shoulder rotational peak torque relative to body mass?
* Does WJR influence the external/internal shoulder rotation ratio in dominant and non-dominant arms at varying angular velocities? Researchers will compare pre- and post-intervention isokinetic measurements to see if WJR training leads to significant changes in shoulder strength and balance.

Participants will:

* Incorporate WJR sessions three times per week into their usual CrossFit training.
* Undergo isokinetic testing of both shoulders at baseline and post-intervention at 60°/s, 180°/s, and 300°/s.
* Have their training adherence and technique monitored throughout the study.

DETAILED DESCRIPTION:
Model: Single Group

Model Description:

This study followed a single-arm, quasi-experimental pre-post design in which all participants underwent the same intervention: six weeks of weighted jump rope (WJR) training, integrated into their regular CrossFit routines. The intervention's impact on isokinetic shoulder strength variables was assessed by comparing pre- and post-intervention measures within the same group of participants.

Number of Arms

1, Only one group received the intervention-there was no control or comparator group.

Masking Outcomes Assessor.

Masking Description:

Due to the nature of the physical intervention (WJR training), blinding participants and care providers was not feasible. However, outcome assessors conducting the isokinetic tests were blinded to the study's hypotheses and group allocations to reduce measurement bias.

Allocation N/A. Participants were not randomly assigned but instead enrolled in a single group to undergo the same intervention protocol.

Enrollment 18 participants

ELIGIBILITY:
Inclusion Criteria:

* self-reported CrossFit training experience. Accordingly, participants were classified into one of three categories (Torres-Banduc et al., 2021): advanced level (≥36 months of regular training, defined as ≥3 sessions of ≥120 minutes per week); intermediate level (12 to <36 months); and beginner level (6 to <12 months).
* no injuries in the three months preceding the study.

Exclusion Criteria:

* musculoskeletal issues impacting muscle strength or the ability to undergo isokinetic shoulder evaluation.
* self-reported use of anabolic steroids or other prohibited substances that might influence the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Rotational peak torque relative to body mass | From enrollment to the end of wieghted jump rope training protocol at 6 weeks
  This variable represents the highest muscular force produced during a shoulder rotation movement, normalized to the participant's body mass (expressed in Nm/kg). It was measured using an isokinetic dynamometer, which quantifies muscle torque under controlled speed and resistance conditions. Participants performed maximal effort shoulder rotations to the left and right at a standardized angular velocity, with proper stabilization to isolate shoulder movement. Normalizing torque to body mass allows comparisons between individuals of different sizes and helps assess the relative strength of the shoulder rotator muscles. Higher values indicate greater rotational strength relative to body weight, which is important for upper limb performance and injury prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano A. Torres-Banduc, PhD., Principal Investigator — University of Americas
Locations (1):
- Human Movement Analysis Laboratory, Viña del Mar, V región/Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be publicly shared, but may be made available upon reasonable request to the corresponding author. This approach ensures data privacy and confidentiality, while still allowing access for valid scientific purposes.

REFERENCES:
- [Background] Torres-Banduc MA, Jerez-Mayorga D, Moran J, Keogh JWL, Ramirez-Campillo R. Isokinetic force-power profile of the shoulder joint in males participating in CrossFit training and competing at different levels. PeerJ. 2021 Sep 17;9:e11643. doi: 10.7717/peerj.11643. eCollection 2021. PMID 34616590
- [Background] Duzgun I, Baltaci G, Colakoglu F, Tunay VB, Ozer D. The effects of jump-rope training on shoulder isokinetic strength in adolescent volleyball players. J Sport Rehabil. 2010 May;19(2):184-99. doi: 10.1123/jsr.19.2.184. PMID 20543219
- [Derived] Torres-Banduc MA, Thapa RK, Perez MA, Ramirez-Campillo R. Isokinetic shoulder strength adaptations to weighted jump rope training in CrossFit athletes: A pre-post study. Shoulder Elbow. 2025 Dec 30:17585732251409407. doi: 10.1177/17585732251409407. Online ahead of print. PMID 41479676